CLINICAL TRIAL: NCT00482690
Title: Analysis of Aldehyde Biomarkers of Exposure and Host Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: primary analyses found unfeasible
Sponsor: University of Nebraska (Other)
Collaborators: R.J. Reynolds Tobacco Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0257-05-FB
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Biomarkers; Aldehydes; Exhaled breath; Harm Reduction; Cigarette smoking; cessation; reduction
MeSH Terms: conditions — Smoking Cessation; Harm Reduction; Cigarette Smoking | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Chewing Gum; Transdermal Patch; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine replacement therapy (NRT) (Experimental): open label NRT self comparator design
  Interventions: Drug: nicotine polacrilex; Drug: nicotine transdermal system; Drug: nicotine inhaler

INTERVENTIONS:
Drug: nicotine polacrilex
  Other Names: Nicorette, gum, lozenge
Drug: nicotine transdermal system
  Other Names: patch
Drug: nicotine inhaler
  Other Names: Nicorette inhaler

SUMMARY:
Analysis of aldeyde biomarkers of exposure and host response The purpose of this prospective, open-label, clinical trial is to establish the feasibility and validity of exhaled breath condensate (EBC) biomarkers for use in studies designed to evaluate harm reduction strategies of smoking. This will be accomplished by measuring selected markers in EBC believed related to the pathogenesis of lung disease before and after a smoking cessation intervention.

DETAILED DESCRIPTION:
Twenty subjects will be accrued in three groups based on smoking habit: 10-20, 20-30 and >30 cigarettes/day. Eligibility criteria include male and female cigarette smokers ≥19 years of age, who are able to give informed consent, able to exhale into Eco Screen instrument for 15-20 minutes. All must be willing to make a serious quit attempt and be willing to use nicotine replacement therapy.

Subjects will be excluded if any of the following are present: regular use of anti-inflammatory medication; presence of any inflammatory disease of the respiratory tract including moderate or worse COPD (FEV1 < 80% predicted and FEV1/FVC ratio < 0.7). Subjects with normal lung function who meet criteria for diagnosis of chronic bronchitis will be excluded. Subjects with stable medical conditions, excluding inflammatory lung disease, will be permitted to participate, providing anti-inflammatory therapies are not used regularly and providing there has been no change in their clinical status in the two months prior to beginning the study.

Upon entering into the study, subjects will establish a quit date and will be treated with nicotine replacement therapy (NRT) products based on individual preference and will receive smoking cessation counseling. They will then be seen at 12 visits over the course of 25 weeks.

Evaluations will include vital signs, interval smoking history, food frequency questionnaire, exhaled carbon monoxide, blood drawn for chemistry and CBC, peripheral blood harvested and serum aliquoted and saved for future biochemical analysis, urine sample for isoprostane, pregnancy test for females, and exhaled breath condensate. Some visits may also include spirometry with and with out bronchodilators, 24 hour urine collections for NNAL and NNAL-glc quantification, health status assessed using St. George's Respiratory Questionnaire, the Functional Assessment of Chronic Illness Therapy - Fatigue, the Leicester Cough Questionnaire, the Clinical COPD Questionnaire and smoking related symptoms assessed using the Breathlessness, Cough, and Sputum Scale.

ELIGIBILITY:
Inclusion Criteria:

* Smokers of at least 5 pack years;
* Stable smoking habit for 3 months;
* Willing to make a serious quit attempt;
* Able to use nicotine replacement therapy

Exclusion Criteria:

* Regular use of anti-inflammatory medication
* Inflammatory lung disease
* Unstable medical condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-08-23 (Actual); Primary Completion 2007-09-09 (Actual); Study Completion 2007-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I Rennard, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Replacement Therapy Open Label: open label NRT self comparator design
  nicotine polacrilex
  nicotine transdermal system
  nicotine inhaler
Period: Overall Study
Arm/Group | Nicotine Replacement Therapy Open Label
Started | 35
Completed | 17
Not Completed | 18

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Replacement Therapy: open label NRT self comparator design
  nicotine polacrilex
  nicotine transdermal system
  nicotine inhaler
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Study conducted exclusively in Omaha NE
  participants
    United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Aldehyde Biomarkers
Description: Aledhydes were assessed in exhaled breath condensate by mass spec and chemical assay.
Time Frame: Study was terminated at an interim analysis for futility
Population: no data were analyzed as specimen collection was inadequate for analysis
Arm/Group | Nicotine Replacement Therapy Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Nicotine Replacement Therapy Open Label
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No